CLINICAL TRIAL: NCT01020799
Title: A Phase II, Multi-center, Randomized, Double-bind, Double-dummy, Active and Placebo Controlled, Parallel Group Study to Assess the Efficacy and Safety of AZD7268 in Patients With Major Depressive Disorder
Brief Title: AZD7268 Safety and Tolerability Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1151C00005
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD7268 (Experimental): The AZD7268 15 mg BID arm consisted of 3 AZD7268 5 mg capsules dosed orally in the morning and evening. In addition, 2 placebo tablets to match encapsulated escitalopram tablets were dosed orally in the morning only.
  Interventions: Drug: AZD7268; Drug: Placebo tablets
- Placebo (Placebo Comparator): The placebo arm consisted of 3 placebo capsules to match AZD7268 capsules dosed orally in the morning and evening. In addition, 2 placebos to match encapsulated escitalopram tablets were dosed orally in the morning only.
  Interventions: Drug: Placebo capsules; Drug: Placebo tablets
- Escitalopram (Active Comparator): The escitalopram 20 mg QD arm consisted of 3 placebo to match AZD7268 capsules dosed orally in the morning and evening. In addition, during Week 1, one encapsulated 10-mg escitalopram tablet and 1 placebo to match encapsulated escitalopram tablet were dosed orally in the morning only. During Weeks 2 through 4, two encapsulated 10-mg escitalopram tablets were dosed orally in the morning only.
  Interventions: Drug: Escitalopram; Drug: Placebo capsules

INTERVENTIONS:
Drug: AZD7268 — 15 mg, oral, twice daily (BID)
  Arms: AZD7268
Drug: Escitalopram — 20 mg, oral, once daily (QD)
  Arms: Escitalopram
Drug: Placebo capsules — Placebo capsules to match AZD7268
  Arms: Escitalopram; Placebo
Drug: Placebo tablets — Placebo tablets to match encapsulated escitalopram
  Arms: AZD7268; Placebo

SUMMARY:
The purpose of this study is to prove the principle that treatment with AZD7268 reduces depressive symptoms in patients with Major Depressive Disorder (MDD) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written, and dated Informed Consent prior to any study specific procedures
* Documented primary clinical diagnosis meeting criteria from the DSM-IV, Text Revision (APA 2000) for any of the following:
* 296.2x Major Depressive Disorder, Single Episode, or
* 296.3x Major Depressive Disorder, Recurrent

Exclusion Criteria:

* Patients with a secondary DSM-IV Axis I disorder other than GAD or social anxiety disorder (as assessed by MINI), provided the primary diagnosis is MDD. This diagnosis should have been made at least 6 months before enrollment
* Patients with a diagnosis of DSM-IV Axis II disorder which has a major impact on the patient's current psychiatric status
* Patients whose current episode of depression started less than 4 weeks before enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Research Site, Birmingham, Alabama
  - Research Site, Garden Grove, California
  - Research Site, San Diego, California
  - Research Site, New Haven, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Rockville, Maryland
  - Research Site, Cedarhurst, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Dayton, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Memphis, Tennessee
  - Research Site, Friendswood, Texas
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 centers were inititated with first patient enrolled on 16 November 2009 and last patient completed on 15 April 2010. A total of 430 patients were enrolled with 247 qualified patients allocated to randomized treatment.
Pre-assignment Details: Patients were required to discontinue current treatment for MDD at least 7 days prior to randomization (14 days prior to Day 1 for monoamine oxidase inhibitors [MAOIs] and 28 days prior to Day 1 for fluoxetine). Patients not taking medications for MDD at enrollment could be randomized once eligibility was confirmed.
Groups:
- AZD7268: AZD7268 15 mg twice per day (BID), placebo matching escitalopram
- Placebo: Placebo matching both AZD7268 and escitalopram
- Escitalopram: Escitalopram 20 mg once per day(QD) Placebo matching AZD7268
Period: Overall Study
Arm/Group | AZD7268 | Placebo | Escitalopram
Started | 98 | 99 | 50
Patients Received Treatment | 96 | 99 | 50
Full Analysis Set | 91 | 94 | 49
Completed | 79 | 85 | 43
Not Completed | 19 | 14 | 7
Not completed — Adverse Event | 4 | 3 | 2
Not completed — non-compliance; lack of efficacy; etc. | 4 | 3 | 0
Not completed — Protocol Violation | 3 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Lost to Follow-up | 6 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7268 | Placebo | Escitalopram | Total
Number analyzed (Participants) | 98 | 99 | 50 | 247
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.29 (11.63) | 41.77 (10.02) | 36.22 (11.29) | 39.09 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 49 | 22 | 108
  Male | 61 | 50 | 28 | 139
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 66 | 56 | 34 | 156
  Black or African American | 27 | 35 | 15 | 77
  Asian | 0 | 4 | 1 | 5
  Native Hawaiian or other Pacific Islander | 1 | 1 | 0 | 2
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Other | 3 | 3 | 0 | 6
Montgomery-Åsberg Depression Rating Scale (MADRS) total score at baseline [Mean (Standard Deviation); unit: scores on a scale] — MADRS total score, sum of 10 item scores (each on a 0 (best value) to 6 (worst value)scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 60 (the worst). [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
  scores on a scale | 30.9 (3.9) | 31.4 (4.2) | 30.8 (4.0) | 31.03 (4.03)
Hamilton Rating Scale for Depression (HAM-D) total score at baseline [Mean (Standard Deviation); unit: scores on a scale] — HAM-D total score, sum of 17 item scores (each on a 0 to 2 or 0 to 4 scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 52 (the worst). [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
  scores on a scale | 24.3 (2.9) | 24.6 (2.8) | 24.4 (2.8) | 24.43 (2.83)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score Change From Baseline to Week 4.
Description: MADRS total score, sum of 10 item scores (each on a 0 (best value) to 6 (worst value)scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 60 (the worst). Change from baseline was calculated as Week 4 value minus baseline value. [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
scores on a scale | -11.78 (1.13) [lower limit 1.13] | -11.45 (1.05) [lower limit 1.05] | -11.70 (1.57) [lower limit 1.57]

2. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Response
Description: Number of patients with MADRS response at Week 4. MADRS response is defined as >=50% reduction in MADRS total score from baseline. MADRS total score, sum of 10 item scores (each on a 0 (best value) to 6 (worst value)scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 60 (the worst). MADRS response at Week 4 is calculated using last observation carried forward (LOCF). [Full Analysis Set (FAS)]
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
Participants | 31 | 31 | 14

3. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Remission
Description: Number of patients, who achieved MADRS remission at week 4. Remission is defined as a MADRS total score <= 10. MADRS total score, sum of 10 item scores (each on a 0 (best value) to 6 (worst value)scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 60 (the worst). MADRS remission at Week 4 is calculated using last observation carried forward (LOCF). [Full Analysis Set (FAS)]
Time Frame: Week 4
Measure: Number; unit: Participants
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
Participants | 20 | 12 | 10

4. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D) Total Score Change From Baseline to Week 4.
Description: HAM-D total score, sum of 17 item scores (each on a 0 to 2 or 0 to 4 scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 52 (the worst). Change from baseline to Week 4 was calculated as Week 4 value minus baseline value. [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
scores on a scale | -9.22 (0.82) [lower limit 0.82] | -9.15 (0.81) [lower limit 0.81] | -9.84 (0.99) [lower limit 0.99]

5. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score Change From Baseline
Description: CGI-S assesses global illness severity, i.e. the patient's current clinical state, on a continuous scale from 1 ("Normal, not ill") to 7 ("Among the most extremely ill patients"). Change from baseline to Week 4 was calculated as Week 4 value minus baseline value. [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
scores on a scale | -1.26 (0.13) [lower limit 0.13] | -1.15 (0.13) [lower limit 0.13] | -1.31 (0.17) [lower limit 0.17]

6. Secondary Outcome: Hamilton Rating Scale for Anxiety (HAM-A) Total Score Change From Baseline
Description: HAM-A total score, sum of 14 item scores (each on a 0 to 4 scale), assesses the severity of anxiety symptoms on a continuous scale from 0 (the best) to 52 (the worst). Change from baseline to Week 4 was calculated as Week 4 value minus baseline value. [observed cases, Mixed Model Repeated Measurement (MMRM), Full Analysis Set (FAS)]
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD7268 | Placebo | Escitalopram
Number analyzed (Participants) | 91 | 94 | 49
scores on a scale | -5.30 (0.60) [lower limit 0.60] | -4.66 (0.61) [lower limit 0.61] | -6.15 (0.78) [lower limit 0.78]

ADVERSE EVENTS:
Arm/Group | AZD7268 | Placebo | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/99 | 0/50
Other Adverse Events (participants affected / at risk) | 36/96 | 33/99 | 26/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7268 (N=96) | Placebo (N=99) | Escitalopram (N=50)
Headache (Nervous system disorders) | 9 | 15 | 7
Fatigue (General disorders) | 5 | 1 | 1
Somnolence (Nervous system disorders) | 4 | 5 | 3
Nasopharyngitis (Infections and infestations) | 3 | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 7
Nausea (Gastrointestinal disorders) | 3 | 4 | 7
Dry Mouth (Gastrointestinal disorders) | 15 | 9 | 3
Libido Decreased (Psychiatric disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation of results until the earlier of the publication of the first multi-center publication and the second anniversary of the completion of the multi-center study at all sites. Sponsor must receive a copy of proposed manuscript for review and comment at least 60 days prior to its submission for publication or presentation.